CLINICAL TRIAL: NCT04929054
Title: Principal Component Regression Based Contrast Enhanced Ultrasound Evaluating System in the Management of BI-RADS 4A Breast Nodules
Brief Title: PCR Based CEUS in BI RADS 4A Nodules
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Breast 2019
Record Dates: First submitted 2021-04-07; First posted 2021-06-18 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-03

CONDITIONS: PCA; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnostic Imaging; In Vitro Meat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pathology results of breast nodules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Diagnostic Test: imaging — ultrasound and contrast enhanced ultrasound for BI RADS4A breast modules
  Other Names: in-vitro

SUMMARY:
The aim of this study was to investigate the added value of Principal Component Regression (PCR) based contrast-enhanced ultrasound (CEUS) for differentiating low risk patients with breast nodules categorized as 4A using the Breast Imaging Reporting and Data System (BI-RADS).

DETAILED DESCRIPTION:
The aim of this study was to investigate the added value of Principal Component Regression (PCR) based contrast-enhanced ultrasound (CEUS) for differentiating low risk patients with breast nodules categorized as 4A using the Breast Imaging Reporting and Data System (BI-RADS). The study included patients with 4A nodules confirmed by core biopsy and/or surgery. The CEUS parameters were assessed and PCR scores were calculated to evaluated the added value in BI-RADS 4A nodules.

ELIGIBILITY:
Inclusion Criteria:

patients with BI-RADS 4A breast lesion

Exclusion Criteria:

(i) absence of a pathologic diagnosis; (ii) presence of breast nodules that were too large to compare with normal parenchyma; (iii) patients with radiotherapy and chemotherapy of breast cancer; and (iv) skin disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with nodules which were sonographically classified as BI-RADS 4 A breast lesion
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
surgery or biopsy | up to 3 months
  According to the PCR result, if it's positive, the nodule category was maintained, however, if it's negative, the nodule was downgraded. all nodules were submitted to biopsy or biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: pintong Huang, Study Chair — SAHZJU
Locations (1):
- SAHZJU, Hanzhou, Zhejiang, China